CLINICAL TRIAL: NCT00104104
Title: A Multicenter,Open Label, Randomized Trial Evaluating the Duration of Infusion of Zoledronic Acid 4 mg IV in Multiple Myeloma Patients With Bone Metastases
Brief Title: A Multiple Myeloma Trial in Patients With Bone Metastases
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CZOL446EUS97; US97
Record Dates: First submitted 2005-02-22; First posted 2005-02-23 (Estimated); Results first posted 2011-06-06 (Estimated); Last update posted 2011-06-29 (Estimated); Status verified 2011-06

CONDITIONS: Multiple Myeloma
Keywords: Z-MAX, multiple myeloma, zoledronic acid, bone metastases
MeSH Terms: conditions — Multiple Myeloma | interventions — Zoledronic Acid

ARMS (2):
- 15 Minute Infusion (Experimental): Participants received 4 mg zoledronic acid intravenously, in 250 mL of fluid, every 3-4 weeks for up to 24 months, over a 15-minute infusion time, but increasing to a 30-minute infusion time if they experienced a clinically relevant rise in serum creatinine that resolved in less than 12 weeks
  Interventions: Drug: zoledronic acid
- 30 Minute Infusion (Experimental): Participants received 4 mg zoledronic acid intravenously, in 250 mL of fluid, every 3-4 weeks for up to 24 months, over a 30-minute infusion time, but increasing to a 45-minute infusion time if they experienced a clinically relevant rise in serum creatinine that resolved in less than 12-weeks.
  Interventions: Drug: zoledronic acid

INTERVENTIONS:
Drug: zoledronic acid — 4 mg zoledronic acid in 250 mL of calcium-free solution (i.e., 0.9% sodium chloride or 5% glucose) administered intravenously.
  Other Names: ZOMETA®

SUMMARY:
The purpose of this trial is to study the safety of treating patients with multiple myeloma and at least one bone lesion with zoledronic acid 4mg intravenously (IV) every 3 - 4 weeks for 2 years. Patients will receive a zoledronic acid infusion for 15 minutes or 30 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older
* Confirmed diagnosis of Multiple Myeloma
* Stable renal function defined as two serum creatinine determinations of < 3 mg/dL
* Calculated creatinine clearance of greater than or equal to 30 mL/min
* ECOG Performance Status of 0 or 1
* Life expectancy of greater than or equal to 9 months
* If the patient is of child-bearing potential, a negative pregnancy test is required at screening, while postmenopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential.
* Ability to comply with trial requirements and give informed consent.

Exclusion Criteria:

* IV Bisphosphonate therapy for more than 3 years.
* Patients with a diagnosis of amyloidosis.
* Known hypersensitivity to zoledronic acid or other bisphosphonates
* Pregnant patients or lactating patients.
* Women of childbearing potential not on a medically recognized form of contraception
* Patients with uncontrolled cardiovascular disease, hypertension, and Type 2 diabetes mellitus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2004-10; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Chair — Novartis Pharmaceuticals
Locations (68):
- United States (68):
  - Hematology Oncology Specialists, Huntsville, Alabama
  - Palo Verde Hematology Oncology, Glendale, Arizona
  - US Oncology, Tucson, Arizona
  - Myeloma Institute For Research Therapy, Little Rock, Arkansas
  - University of Arkansas, Little Rock, Arkansas
  - Pacific Cancer Medical Center, Anaheim, California
  - Comprehensive Blood and Cancer Center, Bakersfield, California
  - Southbay Oncology Hematology Partners, Campbell, California
  - Bay Area Cancer Research Group, Concord, California
  - California Oncology of the Central Valley, Fresno, California
  - Dr. Robert P. Brouillard Inc., La Jolla, California
  - Antelope Valley Cancer Center, Lancaster, California
  - Pacific Shores Medical Group, Long Beach, California
  - North Valley H/O, Mission Hills, California
  - Hematology/Oncology Group of Orange County, Orange, California
  - Desert Hematology Oncology Medical Group, Rancho Mirage, California
  - Camino Medical Group, Sunnyvale, California
  - Oncotherapeutics, West Hollywood, California
  - Greeley Medical Center, Greeley, Colorado
  - Florida Cancer Specialists, Fort Meyers, Florida
  - South Florida Oncology Hematology, Hollywood, Florida
  - Osceola Cancer Center, Kissimmee, Florida
  - Miami Cancer Care, Miami, Florida
  - Pasco Hernado Oncology, New Port Richey, Florida
  - MetCare Oncology, Ormond Beach, Florida
  - Hematology Oncology Associates PA, Pensacola, Florida
  - Hem/Onc Associates of Central Brevard, Rockledge, Florida
  - Augusta Oncology Associates, Augusta, Georgia
  - Georgia Cancer Specialists, Tucker, Georgia
  - Cancer Care Center, New Albany, Indiana
  - Hutchinson Clinic, PA, Hutchinson, Kansas
  - Hematology and Oncology Specialists, New Orleans, Louisiana
  - Maine Center for Cancer Medicine - Blood Disorders, Scarborough, Maine
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - Oncology Hematology Associates, PA, Clinton, Maryland
  - Maryland Oncology-Hematology PA, Columbia, Maryland
  - Hematology Oncology Associates of Ohio & Michigan, Lambertville, Michigan
  - Providence Cancer Center, Clinical Trials Dept, Southfield, Michigan
  - Kansas City Cancer Center, Kansas City, Missouri
  - St. Joseph Oncology, Inc., Saint Joseph, Missouri
  - The Center for Cancer Care and Research, St Louis, Missouri
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Nevada Cancer Center, Las Vegas, Nevada
  - Center for Cancer & Hematology Disease, Cherry Hill, New Jersey
  - Central Jersey Oncology Center, East Brunswick, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - CINJ at Cooper University Hospital, Voorhees Township, New Jersey
  - New Mexico Cancer Care Associates, Santa Fe, New Mexico
  - Hematology Oncology of Western Suffolk, Bay Shore, New York
  - New York Presbyterian Hospital, New York, New York
  - Syracuse Hematology/Oncology PC, Syracuse, New York
  - Dayton Oncology & Hematology, PA, Kettering, Ohio
  - University of Pennsylvania, Philadelphia, Philadelphia, Pennsylvania
  - Pennsylvania Oncology Associates, Philadelphia, Pennsylvania
  - Berks Oncology and Hematology Associates, West Reading, Pennsylvania
  - Hematology & Oncology Associates of RI, Cranston, Rhode Island
  - Roger Williams Hospital Medical Center, Providence, Rhode Island
  - Charleston Hematology Oncology, Charleston, South Carolina
  - Baptist Regional Cancer Center, Knoxville, Tennessee
  - Center for Oncology Research & Treatment, PA, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - Joe Arrington Cancer Research and Treatment Center, Lubbock, Texas
  - Utah Hematology Oncology, Ogden, Utah
  - Oncology Hematology Associates of Southwest VA, Salem, Virginia
  - Western Washington Oncology, Lacey, Washington
  - Swedish Cancer Institute, Seattle, Washington
  - Fox Valley Hematology Oncology SC, Appleton, Wisconsin

REFERENCES:
- See also: Visit NovartisClinicalTrials.com: Pre-qualify for a trial, and view a list of trials and participating study centers. — http://www.novartisclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- 15 - Minute Infusion: Participants received 4 mg zoledronic acid intravenously, in 250 mL of fluid, every 3-4 weeks for up to 24 months, over a 15-minute infusion time, but increasing to a 30-minute infusion time if they experienced a clinically relevant rise in serum creatinine that resolved in less than 12 weeks.
- 30 - Minute Infusion: Participants received 4 mg zoledronic acid intravenously, in 250 mL of fluid, every 3-4 weeks for up to 24 months, over a 30-minute infusion time, but increasing to a 45-minute infusion time if they experienced a clinically relevant rise in serum creatinine that resolved in less than 12-weeks.
Period: Overall Study
Arm/Group | 15 - Minute Infusion | 30 - Minute Infusion
Started | 90 (2 Participants in the 15-minute infusion group did not receive study drug.) | 89 (1 Participants in the 30-minute infusion group did not receive study drug.)
Safety Population (Including Site 74) | 88 | 88
Safety Population (Excluding Site 74) | 85 (Because of GCP violations at Site 74, post-baseline data for 3 patients in this arm were excluded.) | 84 (Because of GCP violations at Site 74, post-baseline data for 4 patients in this arm were excluded.)
Completed | 15 | 17
Not Completed | 75 | 72
Not completed — Adverse Event | 8 | 8
Not completed — Abnormal laboratory value(s) | 20 | 14
Not completed — Lack of Efficacy | 0 | 3
Not completed — Condition no longer requires study drug | 7 | 4
Not completed — Protocol Violation | 5 | 2
Not completed — Withdrawal by Subject | 11 | 15
Not completed — Lost to Follow-up | 3 | 7
Not completed — Administrative problems | 12 | 13
Not completed — Death | 9 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 15 - Minute Infusion | 30 - Minute Infusion | Total
Number analyzed (Participants) | 88 | 88 | 176
Age, Categorical [Count of Participants; unit: Participants] — Demographic data is provided for the entire Safety Population.
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 39 | 47 | 86
    >=65 years | 49 | 41 | 90
Age Continuous [Mean (Standard Deviation); unit: years] | 64.3 (11.95) | 64.0 (11.54) | 64.1 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 39 | 71
  Male | 56 | 49 | 105
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 70 | 69 | 139
  Black | 9 | 13 | 22
  Asian | 1 | 1 | 2
  Other | 8 | 5 | 13
Region of Enrollment [Number; unit: participants]
  United States | 88 | 88 | 176
Time since diagnosis [Mean (Standard Deviation); unit: months] — This baseline measurement was based on n=86, 87.
  months | 12.5 (24.3) | 9.7 (14.1) | 11.1 (19.8)
Calculated creatinine clearance [Mean (Standard Deviation); unit: mL/min] | 87.3 (32.6) | 89.3 (39.5) | 88.3 (36.1)

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants With a Significant Increase in Serum Creatinine at 12 Months
Description: The primary renal safety endpoint was the number of participants with a clinically relevant increase in serum creatinine at 12 months. Serum creatinine was determined prior to each zoledronic acid infusion for all Participants and was considered to be significantly increased if there was an increase of 0.5 mg/dL or more or a doubling of the baseline serum creatinine value.
Time Frame: Baseline and 12 Months
Population: Safety Population: enrolled patients who received at least one dose of study medication, exluding site 74.
Measure: Number; unit: Participants
Arm/Group | 15 - Minute Infusion | 30 - Minute Infusion
Number analyzed (Participants) | 85 | 84
Participants | 17 [0.43 to 2.65] | 13 [0.43 to 2.65]

2. Secondary Outcome: The Number of Participants With a Significant Increase in Serum Creatinine at 24 Months
Description: Serum Creatinine was considered to be significantly increased if there was an increase of 0.5 mg/dL or more or a doubling of the baseline serum creatinine value.
Time Frame: Baseline and 24 Months
Population: Safety Population; enrolled patients who received at least one dose of study medication.
Measure: Number; unit: Participants
Arm/Group | 15 - Minute Infusion | 30 - Minute Infusion
Number analyzed (Participants) | 85 | 84
Participants | 24 [0.53 to 2.13] | 23 [0.53 to 2.13]

3. Secondary Outcome: Time to First Significant Increase in Serum Creatinine
Description: Median time to event in participants who had a clinically relevant increase in serum creatinine.
Time Frame: Up to 24 months
Population: Safety Population; enrolled patients who received at least one dose of study medication. The medians shown are only for patients who had a significant increase by 24 months.
Measure: Median (Full Range); unit: weeks
Arm/Group | 15 - Minute Infusion | 30 - Minute Infusion
Number analyzed (Participants) | 24 | 23
weeks | 21.6 (19.88) [4.1 to 65.0] | 24.4 (31.48) [2.6 to 93.9]

4. Secondary Outcome: Zoledronic Acid Concentrations
Description: Samples for drug concentration analysis were drawn at 10 and 15 minutes into the infusion for participants in the 15-minute infusion group and at 25 and 30 minutes into the infusion for patients in the 30-minute infusion group. The mean and median zoledronic acid concentrations were greater in the 15-minute group than in the 30-minute group at both sampling timepoints.
Time Frame: 24 months
Population: The pharmacokinetic (PK) population was analyzed for zoledronic acid concentration. Participants were considered to be in the PK population if they had evaluable PK data.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 15 - Minute Infusion | 30 - Minute Infusion
Number analyzed (Participants) | 70 | 63
ng/mL
  First Collection (10 minutes, 25 minutes) | 231.1 (185.4) | 186.3 (54.4)
  Second Collection (15 minutes, 30 minutes) | 248.8 (92.0) | 172.0 (48.3)

5. Primary Outcome: The Number of Participants With Disease Progression
Time Frame: 24 Months
Population: Safety Population; enrolled patients who received at least one dose of study medication.
Measure: Number; unit: Participants
Arm/Group | 15 - Minute Infusion | 30 - Minute Infusion
Number analyzed (Participants) | 85 | 84
Participants | 28 | 20

ADVERSE EVENTS:
Description: Because of GCP violations at Site 74, post-baseline data from that site are excluded from analyses, leaving 85 patients in the 15-minute infusion group and 84 patients in the 30-minute infusion group.
Arm/Group | 15 - Minute Infusion | 30 - Minute Infusion
Serious Adverse Events (participants affected / at risk) | 30/85 | 35/84
Other Adverse Events (participants affected / at risk) | 74/85 | 76/84
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 15 - Minute Infusion (N=85) | 30 - Minute Infusion (N=84)
Anaemia (Blood and lymphatic system disorders) | 5 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 4
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 3
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 3 | 1
Atrioventricular block first degree (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 1
Cardiac failure (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 1
Cardio-respiratory arrest (Cardiac disorders) | 1 | 1
Cardiomyopathy (Cardiac disorders) | 1 | 0
Left ventricular hypertrophy (Cardiac disorders) | 1 | 0
Mitral valve disease (Cardiac disorders) | 1 | 0
Mitral valve stenosis (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 1 | 0
Right atrial dilatation (Cardiac disorders) | 1 | 0
Sinus arrhythmia (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0
Subendocardial ischaemia (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 0
Adrenocortical insufficiency acute (Endocrine disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 4
Diverticular perforation (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 1
Faecal incontinence (Gastrointestinal disorders) | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 3
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 3
Asthenia (General disorders) | 4 | 4
Chest discomfort (General disorders) | 2 | 0
Chest pain (General disorders) | 1 | 3
Chills (General disorders) | 0 | 1
Inflammation (General disorders) | 1 | 0
Influenza like illness (General disorders) | 1 | 0
Mucosal inflammation (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 0 | 2
Pain (General disorders) | 1 | 3
Pyrexia (General disorders) | 2 | 3
Suprapubic pain (General disorders) | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 1
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 1
Liver disorder (Hepatobiliary disorders) | 0 | 1
Anaphylactic reaction (Immune system disorders) | 0 | 1
Abdominal abscess (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 2
Bronchitis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 3
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 0 | 1
Meningitis bacterial (Infections and infestations) | 0 | 1
Oral candidiasis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 7 | 2
Pneumonia bacterial (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 2 | 2
Septic shock (Infections and infestations) | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 1
Compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Fractured sacrum (Injury, poisoning and procedural complications) | 1 | 0
Ilium fracture (Injury, poisoning and procedural complications) | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 3 | 2
Blood bilirubin increased (Investigations) | 0 | 1
Blood calcium abnormal (Investigations) | 1 | 0
Blood creatinine abnormal (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 0 | 1
Blood potassium abnormal (Investigations) | 1 | 0
Blood pressure increased (Investigations) | 1 | 0
Blood urea abnormal (Investigations) | 1 | 0
Brain natriuretic peptide increased (Investigations) | 1 | 0
Ejection fraction abnormal (Investigations) | 1 | 0
Electrocardiogram ST segment elevation (Investigations) | 1 | 0
Hepatic enzyme increased (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 1 | 0
Acidosis (Metabolism and nutrition disorders) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 6
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 3 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 2 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 4
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteolysis (Musculoskeletal and connective tissue disorders) | 1 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 4
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Brain oedema (Nervous system disorders) | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 2
Hydrocephalus (Nervous system disorders) | 0 | 1
Lethargy (Nervous system disorders) | 1 | 1
Loss of consciousness (Nervous system disorders) | 0 | 1
Metabolic encephalopathy (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 2 | 2
Confusional state (Psychiatric disorders) | 2 | 0
Depression (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 2
Suicide attempt (Psychiatric disorders) | 1 | 0
Acute prerenal failure (Renal and urinary disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 2 | 2
Renal failure acute (Renal and urinary disorders) | 4 | 0
Renal failure chronic (Renal and urinary disorders) | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 4
Hypotension (Vascular disorders) | 3 | 1
Jugular vein distension (Vascular disorders) | 0 | 1
Jugular vein thrombosis (Vascular disorders) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 15 - Minute Infusion (N=85) | 30 - Minute Infusion (N=84)
Anaemia (Blood and lymphatic system disorders) | 16 | 26
Neutropenia (Blood and lymphatic system disorders) | 6 | 12
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 11
Abdominal pain (Gastrointestinal disorders) | 6 | 5
Constipation (Gastrointestinal disorders) | 20 | 21
Diarrhoea (Gastrointestinal disorders) | 11 | 19
Dyspepsia (Gastrointestinal disorders) | 5 | 5
Nausea (Gastrointestinal disorders) | 16 | 25
Vomiting (Gastrointestinal disorders) | 8 | 12
Asthenia (General disorders) | 5 | 10
Chills (General disorders) | 6 | 7
Fatigue (General disorders) | 30 | 41
Oedema (General disorders) | 5 | 5
Oedema peripheral (General disorders) | 13 | 19
Pain (General disorders) | 6 | 7
Pyrexia (General disorders) | 14 | 16
Bronchitis (Infections and infestations) | 3 | 5
Herpes zoster (Infections and infestations) | 6 | 6
Pneumonia (Infections and infestations) | 5 | 5
Sinusitis (Infections and infestations) | 7 | 8
Upper respiratory tract infection (Infections and infestations) | 13 | 13
Contusion (Injury, poisoning and procedural complications) | 3 | 7
Weight decreased (Investigations) | 6 | 3
Anorexia (Metabolism and nutrition disorders) | 8 | 9
Decreased appetite (Metabolism and nutrition disorders) | 6 | 5
Dehydration (Metabolism and nutrition disorders) | 2 | 5
Hyperglycaemia (Metabolism and nutrition disorders) | 7 | 7
Hypokalaemia (Metabolism and nutrition disorders) | 8 | 13
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 | 16
Back pain (Musculoskeletal and connective tissue disorders) | 17 | 16
Bone pain (Musculoskeletal and connective tissue disorders) | 10 | 11
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 6
Muscular weakness (Musculoskeletal and connective tissue disorders) | 5 | 7
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 6
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 7 | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 13 | 12
Pain in jaw (Musculoskeletal and connective tissue disorders) | 2 | 5
Dizziness (Nervous system disorders) | 10 | 10
Dysgeusia (Nervous system disorders) | 4 | 6
Headache (Nervous system disorders) | 8 | 8
Hypoaesthesia (Nervous system disorders) | 10 | 3
Neuropathy (Nervous system disorders) | 9 | 6
Neuropathy peripheral (Nervous system disorders) | 7 | 15
Tremor (Nervous system disorders) | 2 | 5
Anxiety (Psychiatric disorders) | 6 | 4
Depression (Psychiatric disorders) | 9 | 5
Insomnia (Psychiatric disorders) | 10 | 14
Cough (Respiratory, thoracic and mediastinal disorders) | 13 | 14
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 | 16
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 7
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 | 5
Rash (Skin and subcutaneous tissue disorders) | 9 | 12
Hot flush (Vascular disorders) | 3 | 6
Hypertension (Vascular disorders) | 2 | 6
Hypotension (Vascular disorders) | 4 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial; or disclosure of the trial results in their entirety.